CLINICAL TRIAL: NCT05746637
Title: Qualitative and Quantitative Study of the Complexity of the Diagnostic Pathway of Children With a Functional Neurological Symptomatology Disorder
Brief Title: The Complexity of the Diagnostic Pathway of Children With a Functional Neurological Symptomatology Disorder
Acronym: TC-HPaS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2021 LEGRAND-VYSKOC
Record Dates: First submitted 2022-11-18; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-12

CONDITIONS: Conversion Disorder in Children
Keywords: adolescents; functional neurological symptom disorder; children; qualitative study
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: The entire study population

SUMMARY:
The goal of this qualitative and quantitative cross-sectional observational study is to describe the complexity of the diagnostic pathway for Functional Neurological Symptomatology Disorder (TSNF) in children and adolescents based on the experience of the different protagonists of care (parents, adolescents, caregivers).

The main question[s] it aims to answer are:

* How do the various stakeholders experiences the care pathway for children and adolescents with a diagnosis of TSNF
* What are their expectations regarding the diagnosis and management of TSNF Participants will be enrolled in interviews in which they will describe their experience. Parents will also answer a lifestyle questionnaire.

DETAILED DESCRIPTION:
Conversion Disorder (CD) or Functional Neurological Symptomatology Disorder (FNSD) is a pathology characterized by the occurrence of non-simulated physical symptoms of neurological appearance in the absence of underlying organic pathology.

The hyperspecialization of medicine makes the therapeutic approach to FNSD very complex for several reasons:

* Pediatric health professionals are trained to diagnose and treat physical disorders and are at a loss when it comes to psychological disorders
* Physicians often increase the number of complementary tests before making a diagnosis of FNSD, for fear of missing a serious or urgent pathology
* Psychiatric diagnosis is a diagnosis of exclusion, and TSNF is therefore often evoked at the end of the treatment, which leads to wandering in the patient's care This delay in diagnosis does not allow patients to receive appropriate care and the consequences can be serious.

The objective of this mixed qualitative and quantitative study is to study the complexity of the care pathway of patients aged 6 to 18 years with a diagnosis of TSNF, as well as their parents and the health professionals who have taken care of them. The collection of their experience will be done by means of semi-structured interviews which will then be analyzed according to the Interpretative Phenomenological Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients

  * Child or adolescent, boy or girl, aged 6 to 17 years inclusive, treated at the Clermont-Ferrand University Hospital for a conversion disorder diagnosed by a psychiatrist during the past year
  * Presence or not of a follow-up in child psychiatry after the diagnosis
  * Agreement of the legal representatives for participation in the study.
  * Affiliation to a Social Security system.
* Parents / legal representatives

  o Adult subject, parent or legal representative of a child or adolescent meeting the above-mentioned inclusion criteria and participating in the study
* Health professionals

  o Person affiliated with the Clermont-Ferrand University Hospital, with experience in caring for children or adolescents with a conversion disorder (pediatrician, psychiatrist, nurse, psychologist,
* For all participants

  * Able to give informed consent to participate in the research.
  * Proficiency in the French language [NB the written language must be mastered by the parents to answer the questionnaires].

Exclusion Criteria:

* For all participants: Present a decompensated somatic or psychiatric pathology or a disorder of vigilance compromising the realization of the research, refusal to participate in the research.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Our population will be a clinical population, made up of children and adolescents aged 6 to 18 years followed at the Clermont-Ferrand University Hospital for TSNF, their parents, and the health professionals who care for them.
  Before the age of 6, it is not easy to talk about oneself and the collection of information is generally done through the parents. After the age of 6, children are able to describe their experience, which allows us to collect their experiences and those of their parents separately. Adolescents between 16 and 18 years of age are often still followed by pediatric teams, and mostly followed by child psychiatry, which justifies the broad cut-off of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Participants' experience of the diagnostic circumstances and care pathway | 1 day
  Obtaining a thematic grid describing the participants' experience of the diagnostic circumstances and care pathway of TSNF in children and adolescents.

SECONDARY OUTCOMES:
Description the diversity of experiences according to each type of participant | 1 day
  Obtaining a thematic grid describing the diversity of experiences according to each type of participant
Participants' expectations regarding the diagnosis and management of TSNF | 1 day
  Obtained a thematic grid describing the participants' expectations regarding the diagnosis and management of TSNF
Total duration of the diagnosis pathway | 1 day
  Total duration (days) between the 1st medical consultation related to TSNF and the 1st psychological consultation (psychiatrist, child psychiatrist, psychologist or multidisciplinary evaluation with psychologist or psychiatrist on the team). This period corresponds to the pre-diagnostic period for the study.
Total number of outpatient consultations related to TSNF | 1 day
  Total number of outpatient consultations related to TSNF during the pre-diagnosis period, including: consultations with general practitioners and specialists other than psychiatrists, consultations in pediatric or adult emergency rooms.
Total number of part-time inpatient stays | 1 day
  Total number of part-time inpatient stays related to TSNF during the pre-diagnosis period
Total number of full-time inpatient stays in the OOH setting | 1 day
  Total number of full-time inpatient stays in the OOH setting during the pre-diagnosis period
Total length of stay in full-time OCM hospitalization | 1 day
  Total length of stay in full-time OCM hospitalization related to TSNF in the pre-diagnosis period.
Presence of one or more biological or radiological additional examination from the list | 1 day
  Presence of at least one biological or radiological additional examination from the following list during the care pathway : biological blood sample, biological cerebrospinal fluid sample, any radiological examination, electroencephalogram or electromyogram related to TSNF or to the search for a differential diagnosis in the pre-diagnostic period.

CONTACTS AND LOCATIONS:
Overall Officials: Aurore Legrand-Viskoc, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France